CLINICAL TRIAL: NCT02185729
Title: Randomized Study Comparing Soybean Oil-Based (Intralipid) With an Olive Oil-Based (ClinOleic) Lipid Emulsion: Effects on Endothelial Function, Inflammatory Markers, Oxidative Stress, Immune Function, Autonomic Nervous System, Insulin Sensitivity and Carbohydrate Metabolism
Brief Title: Comparing Soybean Oil-Based (Intralipid) With an Olive Oil-Based (ClinOleic) Lipid Emulsion on Healthy Volunteers
Acronym: TPN1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00007543
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Diseases, Metabolic; Insulin Sensitivity
Keywords: Intravenous Feeding; Lipid Emulsions, Intravenous
MeSH Terms: conditions — Metabolic Diseases; Insulin Resistance | interventions — soybean oil, phospholipid emulsion; ClinOleic; Glucose; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy Volunteer (Active Comparator): Subjects receive 24 hours of infusion of 0.9% normal saline, dextrose (sugar) without fat, ClinOleic (olive oil-based), and Intralipid (soybean-derived fat)
  Interventions: Drug: Intralipid; Drug: ClinOleic; Drug: Dextrose; Other: Saline (control)

INTERVENTIONS:
Drug: Intralipid — Infusion of Intralipid (soybean-derived fat)
Drug: ClinOleic — Infusion of ClinOleic (olive oil-based)
Drug: Dextrose — Infusion of dextrose (sugar) without fat
Other: Saline (control) — Infusion of 0.9% normal saline

SUMMARY:
Many patients in the hospital who are malnourished or not eating received intravenous feeding or total parenteral nutrition (TPN). Despite improving nutrition, TPN may increase the risk of infections and hospital complications. We do not know why TPN increases hospital complications, but it may be caused by the high sugar or fat content in TPN solutions. The investigators believe that the high sugar and high fat content can limit the ability to fight infections and produce stiffness of blood vessels. This study will compare the effect of high sugar, high fat content or both on blood sugars, blood vessel function, on blood vessel function. The investigators will also compare the effect of different fats (olive oil and soybean) in the TPN solution on the risk of infection and blood vessel function on a total of 12 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, BMI 25 - 35 kg/m2, between the ages of 18 and 65 years

Exclusion Criteria:

* The patient is pregnant or breast feeding
* Subjects have or with history of diabetes, hypertension, fasting triglyceride levels > 250 mg/dL, liver disease (ALT 2.5x > upper limit of normal), serum creatinine ≥1.5 mg/dL
* Smokers or ex-smoker < 3 months of cessation, drug or alcohol abuse
* Mental condition rendering the subject unable to understand the scope and possible consequences of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Siqueira J, Smiley D, Newton C, Le NA, Gosmanov AR, Spiegelman R, Peng L, Osteen SJ, Jones DP, Quyyumi AA, Ziegler TR, Umpierrez GE. Substitution of standard soybean oil with olive oil-based lipid emulsion in parenteral nutrition: comparison of vascular, metabolic, and inflammatory effects. J Clin Endocrinol Metab. 2011 Oct;96(10):3207-16. doi: 10.1210/jc.2011-0480. Epub 2011 Aug 10. PMID 21832112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects seen at Grady Memorial Hospital Clinical Interactions Network unit of the Atlanta Clinical and Translational Science Institute. Subjects were admitted on the afternoon before the study protocol began.
Pre-assignment Details: An overnight fast, subjects underwent research studies in the morning with the infusion starting between 1200 and 1300 h.
Groups:
- Healthy Volunteer: Healthy subjects receive 24-hour TPN infusion of Intralipid (soybean-derived fat), ClinOleic (olive oil), dextrose (sugar) without fat, and a 24-hour infusion of normal saline (control)
  Intralipid
  ClinOleic
  Dextrose
  Saline (control)
Period: 0 Hour (Baseline) of Saline Infusion
Arm/Group | Healthy Volunteer
Started | 12
Completed | 12
Not Completed | 0
Period: 4 Hours Into Saline Infusion
Arm/Group | Healthy Volunteer
Started | 12
Completed | 12
Not Completed | 0
Period: 24 Hours Into Saline Infusion
Arm/Group | Healthy Volunteer
Started | 12
Completed | 12
Not Completed | 0
Period: 0 Hour (Baseline) of Intralipid Infusion
Arm/Group | Healthy Volunteer
Started | 12
Completed | 12
Not Completed | 0
Period: 4 Hours Into Intralipid Infusion
Arm/Group | Healthy Volunteer
Started | 12
Completed | 12
Not Completed | 0
Period: 24 Hours Into Intralipid Infusion
Arm/Group | Healthy Volunteer
Started | 12
Completed | 12
Not Completed | 0
Period: 0 Hour (Baseline) of ClinOleic Infusion
Arm/Group | Healthy Volunteer
Started | 12
Completed | 12
Not Completed | 0
Period: 4 Hours Into ClinOleic Infusion
Arm/Group | Healthy Volunteer
Started | 12
Completed | 12
Not Completed | 0
Period: 24 Hours Into ClinOleic Infusion
Arm/Group | Healthy Volunteer
Started | 12
Completed | 12
Not Completed | 0
Period: 0 Hour (Baseline) of Dextrose Infusion
Arm/Group | Healthy Volunteer
Started | 12
Completed | 12
Not Completed | 0
Period: 4 Hours Into Dextrose Infusion
Arm/Group | Healthy Volunteer
Started | 12
Completed | 12
Not Completed | 0
Period: 24 Hours Into Dextrose Infusion
Arm/Group | Healthy Volunteer
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilation
Description: Endothelium-dependent brachial artery flow-mediated dilation (FMD) was assessed. Ultrasound images of the brachial artery were obtained and arterial diameters were measured with customized software. Brachial artery FMD was calculated as (hyperemic diameter - baseline diameter)/baseline diameter × 100.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: percentage of brachial artery diameter
Groups:
- Intralipid: Healthy subjects receive 24-hour TPN infusion of Intralipid (soybean-derived fat)
- ClinOleic: Healthy subjects receive 24-hour TPN infusion of ClinOleic (olive oil)
- Dextrose: Healthy subjects receive 24-hour TPN infusion of dextrose (sugar) without fat
- Saline: Healthy subjects receive 24-hour infusion of normal saline (control)
Arm/Group | Intralipid | ClinOleic | Dextrose | Saline
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of brachial artery diameter | 10.3 (0.88) | 8.9 (0.80) | 9.2 (0.72) | 9.1 (0.58)

2. Primary Outcome: Flow Mediated Dilation
Description: Endothelium-dependent brachial artery flow-mediated dilation (FMD) was assessed. Ultrasound images of the brachial artery were obtained and arterial diameters were measured with customized software. Brachial artery FMD was calculated as (hyperemic diameter - 4 hour diameter)/4 hour diameter × 100.
Time Frame: 4 hours after infusion
Measure: Mean (Standard Error); unit: percentage of brachial artery diameter
Arm/Group | Intralipid | ClinOleic | Dextrose | Saline
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of brachial artery diameter | 7.9 (0.83) | 9.0 (0.88) | 8.3 (0.67) | 8.2 (1.37)

3. Primary Outcome: Flow Mediated Dilation
Description: Endothelium-dependent brachial artery flow-mediated dilation (FMD) was assessed. Ultrasound images of the brachial artery were obtained and arterial diameters were measured with customized software. Brachial artery FMD was calculated as (hyperemic diameter - 24 hour diameter)/24 hour diameter × 100.
Time Frame: 24 hours after infusion
Measure: Mean (Standard Error); unit: percentage of brachial artery diameter
Arm/Group | Intralipid | ClinOleic | Dextrose | Saline
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of brachial artery diameter | 7.2 (0.74) | 9.1 (0.91) | 10.2 (1.15) | 9.7 (0.89)

ADVERSE EVENTS:
Groups:
- Healthy Volunteer: Healthy subjects receive 24-hour TPN infusion of Intralipid (soybean-derived fat), ClinOleic (olive oil), dextrose (sugar) without fat, and a 24-hour infusion of normal saline (control)
Arm/Group | Healthy Volunteer
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Short duration and involved healthy volunteers--not clear whether the use of olive oil-based lipid emulsions may result in improved clinical outcomes over traditional lipid emulsions in hospitalized patients with medical and surgical illness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No